CLINICAL TRIAL: NCT04145349
Title: A Randomized, Open-Label Phase 1/2 Study Evaluating Ramucirumab in Pediatric Patients and Young Adults With Relapsed, Recurrent, or Refractory Desmoplastic Small Round Cell Tumor
Brief Title: CAMPFIRE: A Study of Ramucirumab (LY3009806) in Children and Young Adults With Desmoplastic Small Round Cell Tumor
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17305; J1S-MC-JV01 (Other: Eli Lilly and Company); 2018-004242-42 (EudraCT Number)
Record Dates: First submitted 2019-10-29; First posted 2019-10-30 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Desmoplastic Small Round Cell Tumor
Keywords: soft tissue sarcoma; adolescents and young adults (AYAs); adolescent
MeSH Terms: conditions — Desmoplastic Small Round Cell Tumor; Sarcoma | interventions — Ramucirumab; Cyclophosphamide; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ramucirumab + Cyclophosphamide + Vinorelbine (Experimental): Participants received the following treatments in a 28-day cycle, continuing until disease progression or a criterion for discontinuation was met.
  * Ramucirumab administered intravenously at a dose of 12 milligrams per kilogram (mg/kg) as a one-hour infusion on days 1 and 15.
  * Cyclophosphamide administered orally at 25 milligrams per meter square (mg/m2) daily from days 1 to 28.
  * Vinorelbine administered intravenously at 25 mg/m² on days 1, 8, and 15.
  Interventions: Drug: Ramucirumab; Drug: Cyclophosphamide; Drug: Vinorelbine
- Cyclophosphamide + Vinorelbine (Active Comparator): Participants received the following treatments in a 28-day cycle, continuing until disease progression or a criterion for discontinuation was met.
  * Cyclophosphamide administered orally at 25 mg/m² daily from days 1 to 28.
  * Vinorelbine administered intravenously at 25 mg/m² on days 1, 8, and 15.
  Interventions: Drug: Cyclophosphamide; Drug: Vinorelbine

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806
  Arms: Ramucirumab + Cyclophosphamide + Vinorelbine
Drug: Cyclophosphamide — Administered orally
Drug: Vinorelbine — Administered IV

SUMMARY:
This study is being conducted to test the safety and efficacy of ramucirumab in combination with other chemotherapy in the treatment of relapsed, recurrent, or refractory desmoplastic small round cell tumor (DSRCT) in children and young adults. This trial is part of the CAMPFIRE master protocol (NCT05999994) which is a platform to accelerate the development of new treatments for pediatric and young adult participants with cancer. Your participation in this trial could last 12 months or longer, depending on how you and your tumor respond.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have discontinued all previous treatments for cancer or investigational agents ≥7 days after the last dose or per the type of previous treatment as stated in the protocol and must have recovered from the acute effects to ≤Grade 2 for alopecia and decreased tendon reflex and to ≤Grade 1 for all other effects at the time of enrollment, unless otherwise noted. Consult with the Lilly clinical research physician or scientist for the appropriate length of time prior to the first dose of study treatment.
* Participants with relapsed, recurrent, or refractory DSRCT.
* Participants must:

  * Have measurable disease by Response Evaluation Criteria in Solid Tumors, Version (RECIST) 1.1.
  * Have received at least one prior line of systemic treatment (including neoadjuvant and adjuvant chemotherapy). This prior treatment must include approved therapies for which they are eligible, unless the participant is not a suitable candidate for the approved therapy.
  * Not be eligible for surgical resection at time of enrollment.
* Adequate cardiac function, defined as: Shortening fraction of ≥27% by echocardiogram, or ejection fraction of ≥50% by gated radionuclide study.
* Adequate blood pressure (BP) control, defined as:

  * Participants ≥18 years: Controlled hypertension defined as systolic BP ≤150 millimeters of mercury (mmHg) or diastolic BP ≤90 mmHg where standard medical management is permitted. Please note that ≥2 serial BP readings should be obtained and averaged to determine baseline BP.
  * Participants <18 years: A BP ≤95th percentile for age, height, and gender measured as described in National High Blood Pressure Education Program Working Group (NHBPEPWG) on High Blood Pressure in Children and Adolescents (2004), where standard medical management is permitted. Please note that ≥2 serial BP readings should be obtained and averaged to determine baseline BP.
* Adequate hematologic function, as defined as:

  * Absolute neutrophil count (ANC): ≥750/microliters (µL) granulocyte-colony stimulating factor (G-CSF) permitted up to 48 hours prior. Participants with documented history of benign ethnic neutropenia or other conditions could be considered with a lower ANC after discussion with and approval from the Lilly clinical research physician or scientist.
  * Platelets: ≥75,000/cubic millimeters. Platelet transfusion permitted up to 72 hours prior.
  * Hemoglobin: ≥8 grams per deciliter (g/dL) (≥80 g/liter). Transfusions to increase the participant's hemoglobin level to at least 8 g/dL are permitted; however, study treatment must not begin until 7 days after the transfusion, and complete blood count criteria for eligibility are confirmed within 24 hr of first study dose.
* Adequate renal function, as defined as:

  * Creatinine clearance or radioscope glomerular filtration rate (GFR) ≥60 milliliters/minute/meters squared OR serum creatinine meeting the following parameters:

    * for participants ≥18 years of age serum creatinine ≤1.5×upper limit of normal (ULN);
    * for participants <18 years of age, serum creatinine based on age/gender as follows: Age 1 to <2 years maximum serum creatinine 0.6, Age 2 to <6 years maximum serum creatinine 0.8, Age 6 to <10 years maximum serum creatinine 1.0, Age 10 to <13 years maximum serum creatinine 1.2, Age 13 to <16 years maximum serum creatinine 1.5 for males and 1.4 for females, Age 16 to <18 years maximum serum creatinine 1.7 for males and 1.4 for females.
  * Urine protein meeting the following parameters:

    * for participants ≥18 years of age: <2+ on dipstick or routine urinalysis. If urine dipstick or routine analysis indicates proteinuria ≥2+, then a 24-hour urine must be collected and must demonstrate <2 grams of protein in 24 hours to allow participation in the study.
    * for participants <18 years of age: ≤30 milligrams per deciliter urine analysis or <2+ on dipstick. If urine dipstick or routine analysis indicates proteinuria ≥2+, then a 24-hour urine must be collected and must demonstrate <1 g of protein in 24 hours to allow participation in the study.
* Adequate liver function:

  * Total bilirubin: ≤1.5×ULN. Except participants with document history of Gilbert Syndrome who must have a total bilirubin level of <3.0×ULN.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST): ≤2.5×ULN OR ≤5.0×ULN if the liver has tumor involvement.
* The participant has an adequate coagulation function as defined by International Normalized Ratio ≤1.5 or prothrombin time ≤1.5×ULN, and partial thromboplastin time ≤1.5×ULN if not receiving anticoagulation therapy. For participants receiving anticoagulants, exceptions to these coagulation parameters are allowed if they are within the intended or expected range for their therapeutic use. Participants must have no history of clinically significant active bleeding (defined as within 14 days of first dose of study drug) or pathological condition that carries a high risk of bleeding (for example, tumor involving major vessels or known esophageal varices).
* The participant has adequate hematologic and organ function ≤1 week (7 days) prior to first dose of study drug.
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to randomization. Male and female participants must agree to use highly effective contraception for the duration of the study and up to 3 months following the last dose of ramucirumab and vinorelbine, and 12 months following the last dose of cyclophosphamide in order to prevent pregnancy.

Exclusion Criteria:

* Participants with severe and/or uncontrolled concurrent medical disease or psychiatric illness/social situation that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol.
* Participants who have active infections requiring therapy.

  * Participants with an active fungal, bacterial, and/or known severe viral infection including, but not limited to, human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required).
* Participants who have had allogeneic bone marrow or solid organ transplant are excluded.
* Surgery: Participants who have had, or are planning to have, the following invasive procedures are not eligible:

  * Major surgical procedure, laparoscopic procedure, or significant traumatic injury within 28 days prior to enrollment.
  * Central line placement or subcutaneous port placement is not considered major surgery.
  * Core biopsy, fine needle aspirate, and bone marrow biopsy/aspirate are not considered major surgeries.
  * Surgical or other wounds must be adequately healed prior to enrollment.
* Bleeding and thrombosis:

  * Participants with evidence of active bleeding or a history of significant (≥Grade 3) bleeding event within 3 months prior to enrollment are not eligible.
  * Participants with a bleeding diathesis or vasculitis are not eligible.
  * Participants with known or prior history in the prior 3 months of esophageal varices are not eligible.
  * Participants with a history of deep vein thrombosis requiring medical intervention (including pulmonary embolism) within 3 months prior to study enrollment are not eligible.
  * Participants with a history of hemoptysis or other signs of pulmonary hemorrhage within 3 months prior to study enrollment are not eligible.
* Cardiac:

  * Participants with a history of central nervous system (CNS) arterial/venous thromboembolic events (VTEs) including transient ischemic attack (TIA) or cerebrovascular accident (CVA) within 6 months prior to study enrollment are not eligible.
  * Participants with myocardial infarction or unstable angina within the prior 6 months.
  * Participants with New York Heart Association Grade 2 or greater congestive heart failure (CHF).
  * Participants with serious and inadequately controlled cardiac arrhythmia.
  * Participants with significant vascular disease (eg, aortic aneurysm, history of aortic dissection).
  * Participants with clinically significant peripheral vascular disease.
* Participants who have a history of fistula, gastrointestinal (GI) ulcer or perforation, or intra-abdominal abscess within 3 months of study enrollment are not eligible.
* Participants with a history of hypertensive crisis or hypertensive encephalopathy within 6 months of study enrollment are not eligible.
* Participants who have non-healing wound, unhealed or incompletely healed fracture, or a compound (open) bone fracture at the time of enrollment are not eligible.
* Participants previously treated and progressed on combination cyclophosphamide and vinorelbine regimen. Participants who received combination as maintenance therapy, without progression, would be eligible.
* Participants with a known hypersensitivity to ramucirumab, cyclophosphamide, vinorelbine or any of the excipients of the medicinal products.
* Hepatic impairment:

  * Severe liver cirrhosis Child-Pugh Class B (or worse).
  * Cirrhosis with a history of hepatic encephalopathy.
  * Clinically meaningful ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis.
  * History of hepatorenal syndrome.
* The participant has a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (eg, hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
* The participant has a urinary outflow obstruction.
* The participant has Grade 2 hematuria or non-infectious cystitis at the time of screening.
* Participants with central nervous system (CNS) involvement are ineligible.

Ages: 12 Months to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2026-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- United States (6):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
- Royal Children's Hospital, Parkville, Victoria, Australia
- Germany (3):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Humanitas, Rozzano, Milano
  - Ospedale Pediatrico Bambino Gesù, Rome, Roma
  - Azienda Ospedaliera di Padova, Padua, Veneto
- Japan (2):
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitario Virgen Del Rocio, Seville
- United Kingdom (4):
  - University College London Hospital, London, London, City of
  - Royal Marsden Hospital (Sutton), London, Sutton
  - Royal Manchester Children's Hospital, Manchester
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: CAMFIRE: A Study of Ramucirumab (LY3009806) in Children and Young Adults With Desmoplastic Small Round Cell Tumor — https://trials.lilly.com/en-US/trial/227439

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ramucirumab + Cyclophosphamide + Vinorelbine | Cyclophosphamide + Vinorelbine
Started | 20 | 10
Received at Least One Dose of Study Drug | 20 | 10
Completed (Completers included participants who died due to any cause or were alive and on study at conclusion but off treatment.) | 17 | 8
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — On study treatment (Ongoing) | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Ramucirumab + Cyclophosphamide + Vinorelbine: Participants received the following treatments in a 28-day cycle, continuing until disease progression or a criterion for discontinuation was met.
  * Ramucirumab administered intravenously at a dose of 12 mg/kg as a one-hour infusion on days 1 and 15.
  * Cyclophosphamide administered orally at 25 mg/m² daily from days 1 to 28.
  * Vinorelbine administered intravenously at 25 mg/m² on days 1, 8, and 15.
- Total: Total of all reporting groups
Arm/Group | Ramucirumab + Cyclophosphamide + Vinorelbine | Cyclophosphamide + Vinorelbine | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.6 (5.67) | 21.4 (5.06) | 20.2 (5.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 15 | 10 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 16 | 8 | 24
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 13 | 4 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9
  Japan | 1 | 3 | 4
  Italy | 3 | 1 | 4
  United Kingdom | 5 | 1 | 6
  Australia | 1 | 0 | 1
  Germany | 3 | 0 | 3
  Spain | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the date of investigator-determined objective progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or death from any cause in the absence of disease progression. Progressive disease (PD) was defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.Participants known to be alive and without disease progression were censored at the date of their last adequate tumor assessment per RECIST 1.1 criteria, or date of randomization (whichever is later). The posterior median and 98% credible interval were estimated using Bayesian analysis. Data are presented as the posterior median with 98% credible interval.
Time Frame: Randomization to Objective Progression or Death Due to Any Cause (Up To 23 Months)
Population: All randomized participants who received at least one dose of study drug (including the censored participants). Number of participants censored in Ramucirumab + Cyclophosphamide + Vinorelbine = 4, Cyclophosphamide + Vinorelbine = 2.
Measure: Median (98% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + Cyclophosphamide + Vinorelbine | Cyclophosphamide + Vinorelbine
Number analyzed (Participants) | 20 | 10
Months | NA [NA to NA] — The posterior median = 5.69, 98% credible interval (3.20 to 10.01) | NA [NA to NA] — The posterior median = 3.73, 98% credible interval (1.76 to 8.29)
Statistical Analysis 1: Comparison: Ramucirumab + Cyclophosphamide + Vinorelbine vs Cyclophosphamide + Vinorelbine; The Bayesian analyses below include posterior mean of Hazard ratio, and credible intervals instead of confidence intervals; Test type: Superiority; Bayesian hierarchical model; Posterior Mean Hazard Ratio = 0.69, 98% CI 2-sided [0.25 to 1.69]; The posterior probability treatment difference is 0.864

2. Secondary Outcome: Overall Response Rate (ORR): Percentage of Participants Who Achieved a Complete Response (CR) or Partial Response (PR)
Description: * The ORR was defined as the percentage of participants achieving either a CR or PR. Tumor response was assessed based on histology: Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) was used for solid tumors, and Response Assessment in Neuro-Oncology criteria were used for glioblastoma.
  * CR was defined as the disappearance of all target lesions, with any pathological lymph nodes (whether target or non-target) showing a reduction in the short axis to <10 mm. Tumor marker results were required to have normalized. PR was defined as a decrease of at least 30% in the sum of the diameters of target lesions, using baseline diameters as the reference.
Time Frame: Randomization until measured progressive disease (Up To 23 Months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Ramucirumab + Cyclophosphamide + Vinorelbine | Cyclophosphamide + Vinorelbine
Number analyzed (Participants) | 20 | 10
Percentage of participants | 10 [2.7 to 24.5] | 10 [1.1 to 33.7]

3. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the date that measurement criteria for CR or PR (whichever is first recorded) are first met until the first date that disease is recurrent or objective disease progression is observed, per RECIST 1.1 criteria, or the date of death from any cause in the absence of documented disease progression or recurrence .Participants known to be alive and without disease progression were censored at the date of their last adequate tumor assessment per RECIST 1.1 criteria, or date of randomization (whichever is later).
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up To 23 Months)
Population: All randomized participants who received at least one dose of study drug and who had CR or PR responses (including the censored participants). Number of participants censored in Ramucirumab + Cyclophosphamide + Vinorelbine = 0, Cyclophosphamide + Vinorelbine = 1.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + Cyclophosphamide + Vinorelbine | Cyclophosphamide + Vinorelbine
Number analyzed (Participants) | 2 | 1
Months | 9.55 [4.89 to NA] — There were not enough events to estimate the upper limit of the 80% confidence interval. | NA [NA to NA] — Estimation of the median and the 80% confidence interval limits (lower and upper) was not possible as the participant did not achieve the event and was censored.

4. Secondary Outcome: Complete Response (CR) : Percentage of Participants Who Achieved a CR
Description: CR was defined as the disappearance of all target lesions, with any pathological lymph nodes (whether target or non-target) showing a reduction in the short axis to <10 mm.Tumor marker results were required to have normalized.
Time Frame: Randomization until measured progressive disease (Up To 23 Months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Ramucirumab + Cyclophosphamide + Vinorelbine | Cyclophosphamide + Vinorelbine
Number analyzed (Participants) | 20 | 10
Percentage of participants | 5.0 [0.5 to 18.1] | 0 [0.0 to 20.6]

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration of Ramucirumab (Cmax)
Description: Cmax was the concentration of study drug in the blood after the dose is administered. It was measured post-dose and was summarized using descriptive statistics.
Time Frame: End of ramucirumab infusion on Day 1 of Cycle 1
Population: All randomized participants who received at least one dose of Ramucirumab and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Ramucirumab + Cyclophosphamide + Vinorelbine
Number analyzed (Participants) | 14
microgram per milliliter (µg/mL) | 238 (35)

6. Secondary Outcome: PK: Minimum Serum Concentration of Ramucirumab (Cmin)
Description: Cmin was the concentration of study drug in the blood immediately before the next dose was administered. It was measured pre-dose at all visits and was summarized using descriptive statistics.
Time Frame: Prior to ramucirumab infusion on - Day 15 of Cycle 1 and Day 1 of Cycles 2, 4, 7, and 10
Population: All randomized participants who received at least one dose of Ramucirumab and had evaluable PK data for this outcome. Number analyzed refers to participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Ramucirumab + Cyclophosphamide + Vinorelbine
Number analyzed (Participants) | 13
microgram per milliliter (µg/mL)
  Day 15 of Cycle 1 | 41.6 (57)
  Day 1 of Cycle 2: number analyzed (Participants) | 9
  Day 1 of Cycle 2 | 88.7 (47)
  Day 1 of Cycle 4: number analyzed (Participants) | 7
  Day 1 of Cycle 4 | 157 (37)
  Day 1 of Cycle 7: number analyzed (Participants) | 4
  Day 1 of Cycle 7 | 155 (28)
  Day 1 of Cycle 10: number analyzed (Participants) | 2
  Day 1 of Cycle 10 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there were only two participants. Individual values reported:151 µg/mL, 207 µg/mL.

7. Secondary Outcome: Number of Participants With Treatment-Emergent Anti-Drug Antibodies (TE-ADA)
Description: A TE-ADA evaluable participant is considered TE-ADA positive if they have at least one post-baseline ADA titer that is a 4-fold or greater increase from their baseline titer (treatment-boosted); alternatively, if the baseline ADA result is Not Present, the participant is considered TE-ADA positive if there is at least one post-baseline ADA result that is Present with a titer greater than or equal to 1:20 (treatment-induced).
Time Frame: Baseline Up to 23 months
Population: All randomized participants who received at least one dose of study drug and had at least one non-missing baseline, post baseline ADA value.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Cyclophosphamide + Vinorelbine | Cyclophosphamide + Vinorelbine
Number analyzed (Participants) | 13 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline Up to 23 months
Description: * All randomized participants who received at least one dose of study drug. Participants were analyzed based on the actual treatment they received.
  * Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Ramucirumab + Cyclophosphamide + Vinorelbine | Cyclophosphamide + Vinorelbine
All-Cause Mortality (participants affected / at risk) | 12/20 | 7/10
Serious Adverse Events (participants affected / at risk) | 6/20 | 3/10
Other Adverse Events (participants affected / at risk) | 20/20 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Cyclophosphamide + Vinorelbine (N=20) | Cyclophosphamide + Vinorelbine (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Viral diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ramucirumab + Cyclophosphamide + Vinorelbine (N=20) | Cyclophosphamide + Vinorelbine (N=10)
Anaemia (Blood and lymphatic system disorders) | 8 (13) | 2 (13)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 11 (28) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 11 (18) | 2 (2)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (7) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (12) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 3 (7)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (11) | 4 (4)
Asthenia (General disorders) | 2 (2) | 2 (4)
Catheter site rash (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (6) | 2 (3)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 4 (4) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (7) | 4 (7)
Thirst (General disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (2) | 0 (0)
Type iv hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Ear lobe infection (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (2) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 1 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3) | 1 (2)
Alanine aminotransferase increased (Investigations) | 10 (15) | 2 (7)
Anion gap decreased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 7 (11) | 2 (7)
Blood alkaline phosphatase increased (Investigations) | 4 (6) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 1 (1)
Blood creatine increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 3 (11) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 2 (6) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (7) | 3 (9)
Neutrophil count decreased (Investigations) | 10 (33) | 5 (22)
Platelet count decreased (Investigations) | 3 (14) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 2 (2)
Weight increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 11 (39) | 6 (26)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (7) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (7) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (12) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (7) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 10 (17) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 9 (14) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1/5 (1) | 0/0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT04145349/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT04145349/SAP_001.pdf